CLINICAL TRIAL: NCT00771888
Title: Open-Label Extension of the LOCKCYST Trial, LOCKCYST: Long Acting Lnareotide as as Volume Reducing Treatment of Polycystic Livers
Brief Title: Open-Label Extension of LOCKCYST Trial
Acronym: LOCKCYST-ext
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Radboud University Nijmegen Medical Center, Radboud University Nijmegen Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL16194.091.07
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Polycystic Liver Disease; Hepatomegaly; Liver Diseases; Polycystic Kidney; Autosomal Dominant
MeSH Terms: conditions — Polycystic liver disease; Hepatomegaly; Liver Diseases; Polycystic Kidney Diseases; Multiple Pterygium Syndrome, Autosomal Dominant | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): lanreotide
  Interventions: Drug: lanreotide

INTERVENTIONS:
Drug: lanreotide — lanreotide

SUMMARY:
Positive data originating from two polycystic liver patients treated with somatostatin analogues, showed a volume reduction of 38.3% and 14.9%. These two patients had complicated polycystic livers and no other therapeutic options were available.

Patients who participated in LOCKCYST trial are able to benefit from active treatment. Participants will be actively treated for 24 weeks.

DETAILED DESCRIPTION:
van Keimpema L, de Man RA, Drenth JP. Somatostatin analogues reduce liver volume in polycystic liver disease. Gut 2008 September;57(9):1338-9.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the LOCKCYST trial
* 18 yrs-of age
* Multiple cysts > 20
* Cooperating patient
* Is willing and able to comply with the study drug regimen and all other study requirements.
* Willingness to give written informed consent

Exclusion Criteria:

* Use of oral anticonceptives or estrogen suppletion
* Females who are pregnant or breast-feeding
* History or other evidence of chronic pulmonary disease associated with functional limitation
* History of severe cardiac disease (eg, NYHA Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases). In addition, patients with documented or presumed coronary artery disease or cerebrovascular disease should not be enrolled.
* History or other evidence of severe illness or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Symptomatic gallstones (lanreotide decreases gall bladder volume)
* Renal failure requiring hemodialysis

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Liver volume reduction | 24 weeks

SECONDARY OUTCOMES:
Kidney volume Cyst volume | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joost PH Drenth, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; Frederik Nevens, MD, PhD, Principal Investigator — University Hospital Gasthuisberg, University of Leuven; Loes van Keimpema, MSc, Principal Investigator — Radboud University Nijmegen Medical Center
Locations (2):
- University Hospital Gasthuisberg, University of Leuven, Leuven, Belgium
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] van Keimpema L, de Man RA, Drenth JP. Somatostatin analogues reduce liver volume in polycystic liver disease. Gut. 2008 Sep;57(9):1338-9. doi: 10.1136/gut.2008.155721. No abstract available. PMID 18719151